CLINICAL TRIAL: NCT00723736
Title: Non-Interventional Study of the Safe Use of Aerius in Pediatric Patients With Allergic Rhinitis or Chronic Idiopathic Urticaria.
Brief Title: Safety of Aerius Syrup in Pediatric Patients Aged 1-5 Years Old With Allergic Rhinitis or Chronic Idiopathic Urticaria (Study P04446AM1)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P04446
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2009-08-06 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis; Urticaria
MeSH Terms: conditions — Rhinitis; Urticaria | interventions — desloratadine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Patients: Those with allergic rhinitis or chronic idiopathic urticaria.
  Interventions: Drug: Desloratadine

INTERVENTIONS:
Drug: Desloratadine — 2.5 ml (1.25 mg) once daily
  Other Names: Aerius; SCH 034117

SUMMARY:
The objective of this non-interventional study is to evaluate the safety of Aerius syrup in pediatric patients aged 1-5 years old with allergic rhinitis or chronic idiopathic uticaria. The patients will receive 2.5 ml (1.25 mg) once daily.

DETAILED DESCRIPTION:
Pediatric patients aged 1-5 years

ELIGIBILITY:
Inclusion Criteria:

* Patients with allergic rhinitis or chronic idiopathic urticaria
* Aged 1-5 years old
* Caregiver's consent to participate

Exclusion Criteria:

* Healthy individuals
* Younger or older than the 1-5 year old age range

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric clinics around Hungary.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Aerius® Syrup: Aerius® (SCH 34117, desloratadine, DL) syrup administered to those with allergic rhinitis or chronic idiopathic urticaria
Period: Overall Study
Arm/Group | Aerius® Syrup
Started | 100
Completed | 99 (Subject's caregiver did not wish to continue, reasons unrelated.)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aerius® Syrup
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.1 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 55

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Adverse Events
Description: An adverse event is any untoward medical occurrence or unfavorable and unintended sign in a subject administered a pharmaceutical product, whether or not considered related to the use of that product. This includes the onset of new illness and the exacerbation of pre-existing conditions.
Time Frame: Follow-up visit at 3 - 5 weeks after treatment initiation
Measure: Number; unit: participants
Arm/Group | Aerius® Syrup
Number analyzed (Participants) | 100
participants
  Gastrointestinal Disorders | 20
  General Disorders & Administration Site Conditions | 4
  Infections and Infestations | 21
  Respiratory, Thoracic, and Mediastinal Disorders | 6
  Skin and Subcutaneous Tissue Disorders | 4

ADVERSE EVENTS:
Arm/Group | Aerius® Syrup
Serious Adverse Events (participants affected / at risk) | 1/100
Other Adverse Events (participants affected / at risk) | 6/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerius® Syrup (N=100)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerius® Syrup (N=100)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any trial related information may be released by the PI to third party only after written consent is obtained from the sponsor. This restriction is valid until 5 years after study closure.